CLINICAL TRIAL: NCT00590863
Title: Combining Medications to Enhance Depression Outcomes
Acronym: CO-MED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N01 MH090003-02; DSIR AT (Registry Identifier: NCT00590863); N01MH090003 (NIH)
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Major Depressive Disorder
Keywords: depression, medication, antidepressant, chronic, recurrent
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Bronchiolitis Obliterans Syndrome; Recurrence | interventions — Selective Serotonin Reuptake Inhibitors; Escitalopram; Mirtazapine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SSRI + placebo (Active Comparator): Participants will take escitalopram plus placebo.
  Interventions: Drug: SSRI + placebo
- Escitalopram + Bupropion SR (Active Comparator): Participants will take escitalopram + bupropion-SR.
  Interventions: Drug: Escitalopram + Bupropion SR
- Venlafaxine XR + Mirtazapine (Active Comparator): Participants will take venlafaxine-XR + mirtazapine.
  Interventions: Drug: Venlafaxine XR + Mirtazapine

INTERVENTIONS:
Drug: SSRI + placebo — Participants will take escitalopram (10 - 20 mg/day)+ placebo (1 to 3 pills per day). Medications taken orally. Participants will take escitalopram plus placebo for up to 28 weeks. Dosages were adjusted as need at each clinic visit.
  Other Names: escitalopram; placebo
  Arms: SSRI + placebo
Drug: Escitalopram + Bupropion SR — Participant will take Burpopion SR (150 to 450 mg/day) + Escitalopram (10 to 20 mg/day) for up to 28 weeks. Medications taken orally. Bupropion SR was blinded, and escitalopram was given open label. Dosages were adjusted as need at each clinic visit.
  Other Names: escitalopram; bupropion-SR
  Arms: Escitalopram + Bupropion SR
Drug: Venlafaxine XR + Mirtazapine — Participants will take Venlafaxine XR (75 to 225 mg/day) + Mirtazapine (15 to 45 mg/day) for up to 28 weeks. Medications taken orally. Venlafaxine XR was blinded, and mirtazapine was given open label. Dosages were adjusted as need at each clinic visit.
  Other Names: venlafaxine-XR; mirtazapine
  Arms: Venlafaxine XR + Mirtazapine

SUMMARY:
This study will compare whether a combination of antidepressant medications is better than one antidepressant medication alone when given as initial treatment for people with chronic or recurrent major depressive disorder.

DETAILED DESCRIPTION:
The overall aim of Combining Medications to Enhance Depression Outcomes (CO-MED) is to enhance remission rates for outpatients with chronic or recurrent nonpsychotic major depressive disorder (MDD) as defined by DSM-IV TR, treated in primary or psychiatric care settings.

Current evidence indicates that remission, the goal of treatment, is found in only about one-third of representative depressed outpatients treated for up to 14 weeks with an initial SSRI. In addition, even for those who do respond or remit, over one-third relapse in the subsequent 12 months. Combinations of antidepressants are used in practice at the second or subsequent steps when relapse occurs in the longer term, or, in some cases, even acutely as a first step when speed of effect is a clinical priority. Whether such combinations could potentially offer higher remission rates, lower attrition, or greater longer-term benefit if used as initial treatments as compared to monotherapy remains to be examined.

CO-MED will test whether two different medications when given in combination as the first treatment step, compared to one medication, will enhance remission rates, increase speed of remission, be tolerable, and provide better sustained benefits in the longer term. Results of this study will inform practitioners in managing the treatment of patients with chronic or recurrent MDD.

ELIGIBILITY:
Inclusion Criteria:

* Seeking treatment at the primary or specialty care site, and be planning to continue living in the area of that clinic for the duration of the study
* Meets clinical criteria for nonpsychotic MDD, recurrent (with the current episode being at least 2 months in duration), or chronic (current episode greater than 2 years) as defined by a clinical interview and confirmed by the MINI International Neuropsychiatric Interview (MINI)
* Screening 17 item HRSD score of 16 or greater
* Treatment with antidepressant medication combinations is clinically acceptable
* Patient with and without current suicidal ideation may be included in the study as long as outpatient treatment is clinically appropriate

Exclusion Criteria:

* Pregnant or breastfeeding
* Plans to become pregnant over the ensuing 8 months following study entry or are sexually active and not using adequate birth control
* History (lifetime) of psychotic depression, schizophrenia, bipolar (I, II, or NOS), schizoaffective, or other Axis I psychotic disorders
* Current psychotic symptom(s)
* History (within the last 2 years before study entry) of anorexia or bulimia
* Current primary diagnosis of obsessive compulsive disorder
* Current substance dependence that requires inpatient detoxification or inpatient treatment
* Requiring immediate hospitalization for a psychiatric disorder
* Definite history of intolerance or allergy (lifetime) to any protocol medication
* History of clear nonresponse to an adequate trial of an FDA-approved monotherapy in the current MDE if recurrent, or during the last 2 years before study entry if chronic
* History of clear nonresponse to an adequate trial of any study medication used as a monotherapy, or to one or more of the protocol combinations in the current or any prior MDE
* Currently taking any of the study medications at any dose
* Having taken Prozac (fluoxetine) or an MAOI in the 4 weeks before study entry
* Presence of an unstable general medical condition (GMC) that will likely require hospitalization or to be deemed terminal (life expectancy less than 6 months after study entry)
* Currently taking medications or have GMCs that contraindicate any study medications (e.g., seizure disorder)
* Requiring medications for GMCs that contraindicate any study medication
* Epilepsy or other conditions requiring an anticonvulsant
* Lifetime history of having a seizure including febrile or withdrawal seizures
* Receiving or have received vagus nerve stimulation (VNS), electroconvulsive therapy (ECT), repetitive transcranial magnetic stimulation (rTMS), or other somatic antidepressant treatments
* Currently taking or having taken within the 7 days before study entry any of the following exclusionary medications: antipsychotic medications, anticonvulsant medications, mood stabilizers, or central nervous system stimulants (antidepressant medication used for the treatment of depression or other purposes such as smoking cessation or pain are excluded since these agents may interfere with the testing of the major hypotheses under study)
* Uncontrolled narrow angle glaucoma
* Taking thyroid medication for hypothyroidism may be included only if stable on the medication for 3 months
* Using agents within the 7 days before study entry that are potential augmenting agents (e.g., T3 in the absence of thyroid disease, SAMe, St. John's Wort, lithium, buspirone)
* Therapy that is depression-specific

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 665 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar H. Trivedi, MD, Principal Investigator — University of Texas Southwestern Medical Center; Stephen R. Wisniewski, PhD, Study Director — University of Pittsburgh; Diane Warden, PhD, MBA, Study Director — University of Texas Southwestern Medical Center; Kathy Shores-Wilson, PhD, Study Director — University of Texas Southwestern Medical Center; David W. Morris, PhD, Study Director — University of Texas Southwestern Medical Center
Locations (15):
- United States (15):
  - Tuscalossa VA Mental Health Clinic, Tuscaloosa, Alabama
  - Harbor UCLA Family Health Care Center, Harbor City, California
  - UCLA Internal Medicine Clinic, Los Angeles, California
  - Veterans Affairs Medical Center/FIRM Primary Care Clinic, San Diego, California
  - Northwestern Psychiatric Outpatient Treatment Care Center, Chicago, Illinois
  - Clinical Research Institute, Wichita, Kansas
  - MGH/Northshore Medical Center (Salem Psychiatric Facility), Salem, Massachusetts
  - General Psychiatric Ambulatory Clinic, Ann Arbor, Michigan
  - Irving Goldman Primary Care at North Shore Hospital, New York, New York
  - UNC Chapel Hill Adult Diagnostic & Treatment Clinic, Chapel Hill, North Carolina
  - Laureate Psychiatric Clinic and Hospital, Tulsa, Oklahoma
  - Bellefield Clinic of WPIC, Pittsburgh, Pennsylvania
  - Vine Hill Community Clinic, Nashville, Tennessee
  - UT Southwestern Family Medicine Clinic, Dallas, Texas
  - VCU Outpatient Psychiatry Clinic, Richmond, Virginia

REFERENCES:
- [Result] Rush AJ, Trivedi MH, Stewart JW, Nierenberg AA, Fava M, Kurian BT, Warden D, Morris DW, Luther JF, Husain MM, Cook IA, Shelton RC, Lesser IM, Kornstein SG, Wisniewski SR. Combining medications to enhance depression outcomes (CO-MED): acute and long-term outcomes of a single-blind randomized study. Am J Psychiatry. 2011 Jul;168(7):689-701. doi: 10.1176/appi.ajp.2011.10111645. Epub 2011 May 2. PMID 21536692
- [Derived] Olgiati P, Serretti A. Antidepressant emergent mood switch in major depressive disorder: onset, clinical correlates and impact on suicidality. Int Clin Psychopharmacol. 2023 Sep 1;38(5):342-351. doi: 10.1097/YIC.0000000000000479. Epub 2023 Jun 9. PMID 37351585
- [Derived] Olgiati P, Fanelli G, Serretti A. Clinical correlates and prognostic implications of severe suicidal ideation in major depressive disorder. Int Clin Psychopharmacol. 2023 Jul 1;38(4):201-208. doi: 10.1097/YIC.0000000000000461. Epub 2023 Feb 27. PMID 36853754
- [Derived] Olgiati P, Fanelli G, Atti AR, De Ronchi D, Serretti A. Clinical correlates and prognostic impact of binge-eating symptoms in major depressive disorder. Int Clin Psychopharmacol. 2022 Nov 1;37(6):247-254. doi: 10.1097/YIC.0000000000000422. Epub 2022 Jul 12. PMID 35815954
- [Derived] Olgiati P, Serretti A. Persistence of suicidal ideation within acute phase treatment of major depressive disorder: analysis of clinical predictors. Int Clin Psychopharmacol. 2022 Sep 1;37(5):193-200. doi: 10.1097/YIC.0000000000000416. Epub 2022 Jul 7. PMID 35695646
- [Derived] Olgiati P, Fanelli G, Serretti A. Obsessive-compulsive symptoms in major depressive disorder correlate with clinical severity and mixed features. Int Clin Psychopharmacol. 2022 Jul 1;37(4):166-172. doi: 10.1097/YIC.0000000000000396. Epub 2022 Feb 21. PMID 35191860
- [Derived] Olgiati P, Serretti A. Post-traumatic stress disorder and childhood emotional abuse are markers of subthreshold bipolarity and worse treatment outcome in major depressive disorder. Int Clin Psychopharmacol. 2022 Jan 1;37(1):1-8. doi: 10.1097/YIC.0000000000000380. PMID 34686642
- [Derived] Medeiros GC, Prueitt WL, Minhajuddin A, Patel SS, Czysz AH, Furman JL, Mason BL, Rush AJ, Jha MK, Trivedi MH. Childhood maltreatment and impact on clinical features of major depression in adults. Psychiatry Res. 2020 Nov;293:113412. doi: 10.1016/j.psychres.2020.113412. Epub 2020 Aug 18. PMID 32950785
- [Derived] Jha MK, Minhajuddin A, South C, Rush AJ, Trivedi MH. Irritability and Its Clinical Utility in Major Depressive Disorder: Prediction of Individual-Level Acute-Phase Outcomes Using Early Changes in Irritability and Depression Severity. Am J Psychiatry. 2019 May 1;176(5):358-366. doi: 10.1176/appi.ajp.2018.18030355. Epub 2019 Mar 29. PMID 30922100
- [Derived] Sies A, Demyttenaere K, Van Mechelen I. Studying treatment-effect heterogeneity in precision medicine through induced subgroups. J Biopharm Stat. 2019;29(3):491-507. doi: 10.1080/10543406.2019.1579220. Epub 2019 Feb 22. PMID 30794033
- [Derived] De La Garza N, Rush AJ, Killian MO, Grannemann BD, Carmody TJ, Trivedi MH. The Concise Health Risk Tracking Self-Report (CHRT-SR) assessment of suicidality in depressed outpatients: A psychometric evaluation. Depress Anxiety. 2019 Apr;36(4):313-320. doi: 10.1002/da.22855. Epub 2018 Oct 29. PMID 30370613
- [Derived] Gadad BS, Jha MK, Grannemann BD, Mayes TL, Trivedi MH. Proteomics profiling reveals inflammatory biomarkers of antidepressant treatment response: Findings from the CO-MED trial. J Psychiatr Res. 2017 Nov;94:1-6. doi: 10.1016/j.jpsychires.2017.05.012. Epub 2017 May 26. PMID 28628884
- [Derived] Jha MK, Minhajuddin A, Gadad BS, Greer T, Grannemann B, Soyombo A, Mayes TL, Rush AJ, Trivedi MH. Can C-reactive protein inform antidepressant medication selection in depressed outpatients? Findings from the CO-MED trial. Psychoneuroendocrinology. 2017 Apr;78:105-113. doi: 10.1016/j.psyneuen.2017.01.023. Epub 2017 Jan 24. PMID 28187400
- [Derived] Chekroud AM, Zotti RJ, Shehzad Z, Gueorguieva R, Johnson MK, Trivedi MH, Cannon TD, Krystal JH, Corlett PR. Cross-trial prediction of treatment outcome in depression: a machine learning approach. Lancet Psychiatry. 2016 Mar;3(3):243-50. doi: 10.1016/S2215-0366(15)00471-X. Epub 2016 Jan 21. PMID 26803397
- [Derived] Warden D, Trivedi MH, Carmody T, Toups M, Zisook S, Lesser I, Myers A, Kurian KR, Morris D, Rush AJ. Adherence to antidepressant combinations and monotherapy for major depressive disorder: a CO-MED report of measurement-based care. J Psychiatr Pract. 2014 Mar;20(2):118-32. doi: 10.1097/01.pra.0000445246.46424.fe. PMID 24638046
- [Derived] Toups MS, Myers AK, Wisniewski SR, Kurian B, Morris DW, Rush AJ, Fava M, Trivedi MH. Relationship between obesity and depression: characteristics and treatment outcomes with antidepressant medication. Psychosom Med. 2013 Nov-Dec;75(9):863-72. doi: 10.1097/PSY.0000000000000000. Epub 2013 Oct 25. PMID 24163386
- [Derived] Sung SC, Haley CL, Wisniewski SR, Fava M, Nierenberg AA, Warden D, Morris DW, Kurian BT, Trivedi MH, Rush AJ; CO-MED Study Team. The impact of chronic depression on acute and long-term outcomes in a randomized trial comparing selective serotonin reuptake inhibitor monotherapy versus each of 2 different antidepressant medication combinations. J Clin Psychiatry. 2012 Jul;73(7):967-76. doi: 10.4088/JCP.11m07043. Epub 2012 May 29. PMID 22687487
- [Derived] Morris DW, Budhwar N, Husain M, Wisniewski SR, Kurian BT, Luther JF, Kerber K, Rush AJ, Trivedi MH. Depression treatment in patients with general medical conditions: results from the CO-MED trial. Ann Fam Med. 2012 Jan-Feb;10(1):23-33. doi: 10.1370/afm.1316. PMID 22230827
- [Derived] Chan HN, Rush AJ, Nierenberg AA, Trivedi M, Wisniewski SR, Balasubramani GK, Friedman ES, Gaynes BN, Davis L, Morris D, Fava M. Correlates and outcomes of depressed out-patients with greater and fewer anxious symptoms: a CO-MED report. Int J Neuropsychopharmacol. 2012 Nov;15(10):1387-99. doi: 10.1017/S1461145711001660. Epub 2011 Dec 1. PMID 22129562
- [Derived] Zisook S, Lesser IM, Lebowitz B, Rush AJ, Kallenberg G, Wisniewski SR, Nierenberg AA, Fava M, Luther JF, Morris DW, Trivedi MH. Effect of antidepressant medication treatment on suicidal ideation and behavior in a randomized trial: an exploratory report from the Combining Medications to Enhance Depression Outcomes Study. J Clin Psychiatry. 2011 Oct;72(10):1322-32. doi: 10.4088/JCP.10m06724. PMID 22075098

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from March 2008 through April of 2009, with the last subject completing the study in September 2009. Participants were recruited from six primary care and nine psychiatric care sites within the NIMH Depression Trials Network.
Pre-assignment Details: Outpatient enrollees, 18-75 years old, met DSM-IV-TR criteria for either recurrent or chronic MDD. Eligible participants had to be in the index episode for at least two months and to score ≥16 on the 17-item HAM-D. Those with any history of psychotic illness or bipolar disorder, or in need of hospitalization were ineligible.
Groups:
- Escitalopram + Bupropion SR: Participant takes Burpopion SR (150 to 450 mg/day)+ Escitalopram (10 to 20 mg/day) for up to 28 weeks. Medications taken orally. Bupropion SR was blinded, and escitalopram was given open label. Dosages were adjusted as need at each clinic visit.
- Venlafaxine XR + Mirtazapine: Participant takes Venlafaxine XR (75 to 225 mg/day) + Mirtazapine (15 to 45 mg/day) for up to 28 weeks. Medications taken orally. Venlafaxine XR was blinded, and mirtazapine was given open label. Dosages were adjusted as need at each clinic visit.
- Escitalopram + Placebo: Participants will take escitalopram (10 - 20 mg/day)+ placebo (1 to 3 pills per day). Medications taken orally. Participants will take escitalopram plus placebo for up to 28 weeks. Dosages were adjusted as need at each clinic visit.
Period: Overall Study
Arm/Group | Escitalopram + Bupropion SR | Venlafaxine XR + Mirtazapine | Escitalopram + Placebo
Started | 221 | 220 | 224
Completed | 137 | 138 | 146
Not Completed | 84 | 82 | 78

BASELINE CHARACTERISTICS:
Population: Sociodemographic Characteristics
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram + Bupropion SR | Venlafaxine XR + Mirtazapine | Escitalopram + Placebo | Total
Number analyzed (Participants) | 221 | 220 | 224 | 665
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 221 | 220 | 224 | 665
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (13.5) | 42.0 (12.4) | 43.6 (13.1) | 42.7 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 160 | 143 | 452
  Male | 72 | 60 | 81 | 213
Region of Enrollment [Number; unit: participants]
  United States | 221 | 220 | 224 | 665

OUTCOME MEASURES:

1. Primary Outcome: Quick Inventory of Depressive Symptoms
Description: Percentage of patients that achieve remission, as defined as QIDS total score below 6 for last 2 study visits. QIDS depression scores range from 0 (normal) to 27 (very severe).
Time Frame: Measured at Month 7
Population: Remission = Last 2 QIDS < 6. A chi-square test was used to compare the remission rates across the treatment groups. The Fisher's exact test was used when expected cell frequencies were <5. For binary outcomes (e.g., remission), bivariate logistic regression models were fit to estimate the effect of treatment on outcome.
Measure: Number; unit: percentage of participants
Groups:
- Escitalopram + Bupropion SR: Participants will take Escitalopram + BurpopionSR for up to 28 weeks.
- Venlafaxine XR + Mirtazapine: Participants will take Venlafaine XR + Mirtazapine for up to 28 weeks.
- Escitalopram + Placebo: Participants will take escitalopram plus placebo.
  Escitalopram + placebo : Participants will take escitalopram plus placebo for up to 28 weeks.
Arm/Group | Escitalopram + Bupropion SR | Venlafaxine XR + Mirtazapine | Escitalopram + Placebo
Number analyzed (Participants) | 137 | 138 | 146
percentage of participants | 46.6 (5.6) | 41.8 | 46.0 (5.4)

2. Secondary Outcome: Quality of Life Inventory
Description: The Quality of Life Inventory (QOLI) is a 32-item comprehensive self-report of satisfaction in 16 areas of life, such as love, work, and health. Each area is rated in terms of satisfaction and the relationship of that area to overall quality of life. It yields an overall raw score and satisfaction ratings for the 16 individual areas of life. The QOLI raw score is an average of weighted satisfaction ratings computed only over areas of life judged to be Important or Extremely Important to the respondent. Higher scores indicate higher reported quality of life.
Time Frame: Measured at Month 7
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Venlafaxine XR + Mirtazapine: Participants will take Venalfaxine XR + Mirtazapine for up to 28 weeks.
Arm/Group | Escitalopram + Bupropion SR | Venlafaxine XR + Mirtazapine | Escitalopram + Placebo
Number analyzed (Participants) | 137 | 138 | 146
units on a scale | 0.6 (2.1) | 0.4 (2.4) | 0.4 (2.6)

ADVERSE EVENTS:
Description: All potential AEs collected using SAFTEE and FIBSER, but each AE final classification (SAE/OAE) was physicians' decision, and only SAEs were recorded for study. Hence, we are not able to provide complete AE numbers. Please note that all dosing and side effect information is published, and consistent with reported FDA findings and documentation.
Groups:
- Venlafaxine XR + Mirtazapine: Participants will take Venlafaxine XR + Mirtazapine for up to 28 weeks.
- Escitalopram + Placebo: Participants will take Escitalopram + Placebo for up to 28 weeks.
Arm/Group | Escitalopram + Bupropion SR | Venlafaxine XR + Mirtazapine | Escitalopram + Placebo
Serious Adverse Events (participants affected / at risk) | 12/221 | 16/220 | 13/224
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram + Bupropion SR (N=221) | Venlafaxine XR + Mirtazapine (N=220) | Escitalopram + Placebo (N=224)
Death, non-suicide (General disorders) | 0 (0) | 0 (0) | 1 (1)
Medial Hospitialization (Cardiac disorders) | 2 (2) | 5 (5) | 5 (5)
Medical Event, not requiring hospitalizaion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Medical Event, not requiring hospitalization (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Medical Event, not requiring hospitalization (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Medical Event, not requiring hospitalization (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Medical Hospitalization (Surgical and medical procedures) | 1 (1) | 2 (2) | 1 (1)
Medical Hospitalization (General disorders) | 3 (3) | 3 (3) | 3 (3)
Medical Hospitalization (Nervous system disorders) | 3 (3) | 4 (4) | 1 (1)
Medical Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Medical Hospitalization (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Psychiatric Event (non-hospitalized) (Psychiatric disorders) | 1 (1) | 3 (3) | 1 (1)
Psychiatric Hospitalizaion (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Detailed results avaiable. A. J. Rush et al. Combining Medications to Enhance Depression Outcomes (CO-MED): Acute and long-term outcomes: a single-blind randomized study. American Journal of Psychiatry, 2011; 168:689-701.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No